CLINICAL TRIAL: NCT05858853
Title: To Evaluate the Effectiveness of Recombinant Human Serum Albumin Versus Human Serum Albumin in Patients With Hepatic Cirrhosis and Safety of Random, Double-blind, Parallel Grouping Phase II/III Clinical Trial
Brief Title: Phase II/III of Recombinant Human Serum Albumin
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Protgen Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: rHSA 2020-3（Phase Ⅱ）
Record Dates: First submitted 2023-05-05; First posted 2023-05-15 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Hepatic Ascites
MeSH Terms: interventions — recombinant human serum albumin-heme; Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): The experimental drug (recombinant human serum albumin injection) was administered 10 g/ day for 14 days
  Interventions: Drug: Recombinant Human Serum Albumin
- Group 2 (Experimental): The experimental drug (recombinant human serum albumin injection) was administered 20 g/ day for 7 days
  Interventions: Drug: Recombinant Human Serum Albumin
- Group 3 (Active Comparator): Control drug (human blood albumin injection) 10 g/ day for 14 days
  Interventions: Drug: Human serum albumin
- Group 4 (Active Comparator): Control drug (human blood albumin injection) 20 g/ day for 7 days
  Interventions: Drug: Human serum albumin

INTERVENTIONS:
Drug: Recombinant Human Serum Albumin — The experimental drug (recombinant human serum albumin injection) was administered 10 g/ day for 14 days
  Arms: Group 1
Drug: Recombinant Human Serum Albumin — The experimental drug (recombinant human serum albumin injection) was administered 20 g/ day for 7 days
  Arms: Group 2
Drug: Human serum albumin — Control drug (human blood albumin injection) 10 g/ day for 14 days
  Arms: Group 3
Drug: Human serum albumin — Control drug (human blood albumin injection) 20 g/ day for 7 days
  Arms: Group 4

SUMMARY:
This is a randomized, double-blind, position-controlled, parallel group phase II/III clinical study of recombinant human serum albumin (rHSA) in cirrhotic ascites patients.

DETAILED DESCRIPTION:
This is a randomized, double-blind, position-controlled, parallel group phase II/III clinical study of recombinant human serum albumin (rHSA) in cirrhotic ascites patients.

It is divided into two phases: Phase II and Phase III. In phase II, the effect of rHSA on improving serum albumin level in cirrhotic ascites patients will be evaluated with different doses and courses of treatment, and the relationship between dose and efficacy will be determined, so as to provide basis for drug administration plan and sample size calculation of phase III study. In phase III, the efficacy of rHSA will be evaluated with the change of serum albumin concentration from baseline immediately after the completion of the last intravenous administration as the main index, and its safety, PD characteristics and immunogenicity will be further evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Agreed to follow the experimental treatment plan and visit plan, voluntarily enrolled in the group, and signed the informed consent in person;
2. Age ≥18 years old and ≤70 years old, regardless of gender, on the date of signing the informed consent; Body mass index (BMI) was in the range of 18.0 to 29.0 kg/m2 (including boundary values);
3. Patients clinically diagnosed with decompensated cirrhosis with ascites of grade 1 to grade 2 and serum albumin (ALB) <30 g/L were confirmed by abdominal ultrasound examination during the screening period.
4. Fertile men and women of childbearing age (women of childbearing age include premenopausal women and women within 2 years after menopause) are willing to sign the informed consent from the time after the last administration of the investigational drug 3 Take effective contraceptive measures (condom, contraceptive sponge, contraceptive gel, contraceptive film, intrauterine device, oral or injectable contraceptive, subcutaneous implant, etc.) within a month; Pregnancy test results must be negative for women of childbearing age within 7 days or less before the initial trial drug administration.

Exclusion Criteria:

1. People who have a known history of allergy/allergic reaction to yeast or yeast-derived products, or to any component of the study preparation; Allergic constitution (multiple drug or food allergy), or have a history of biological product allergy, other causes Had a history of severe systemic anaphylaxis and was judged by the investigator to be unsuitable for treatment with the experimental drug;
2. At the time of screening, there were severe digestive diseases and complications that were deemed unsuitable for participation in this study by the investigators, including but not limited to malignant ascites and a diagnosis of Grade III or IV liver according to the West-Haven grading criteria Patients with encephalopathy, portal vein cancer thrombus/thrombus, circulatory dysfunction after abdominal puncture, obstructive biliary tract disease identified by ultrasound or other imaging, gastrointestinal bleeding who stopped bleeding less than 10 days after treatment or did not effectively stop bleeding after endoscopic ligation, or who were at greater risk of bleeding during the trial as assessed by the investigator (e.g., before screening) Gastroscopy within 3 months indicated severe esophageal and fundus varices with positive red sign);
3. At the time of screening, there was a history of active cardiovascular disease or other conditions that the investigator judged unsuitable for human albumin therapy, including, but not limited to, hypertension (systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg, The investigators judged that patients were well controlled and stable), severe anemia, acute heart disease, severe cardiopulmonary or structural heart disease, severe arrhythmia, decompensated heart failure (normal or high blood volume), unstable angina, and nearly 6 Myocardial infarction, medicated tachycardia/bradycardia, third-degree atrioventricular block occurred within a month;
4. Patients with active metabolic system diseases or medical history (except diabetic patients with good blood glucose control) at the time of screening, or patients with combined renal function injury who are not suitable for serum albumin treatment according to the investigators;
5. If there are serious underlying diseases during screening, the researchers think it is not suitable to participate in this study. These include, but are not limited to, active malignancies (including hepatocellular carcinoma [HCC]), pulmonary edema, bleeding prone or active bleeding diseases, uncontrolled infections (including active spontaneous bacterial peritonitis [SBP]), thyroid dysfunction (according to the National Cancer Institute Standard for Common Terminology for Adverse Events [NCI CTCAE] version 5.0 3 Grade and above), etc.;
6. The patient has the following abnormalities in laboratory examination:

(1). Liver function: alanine aminotransferase (ALT) > 5×ULN (upper limit of normal value); Aspartate aminotransferase (AST) >5×ULN; Serum bilirubin (TBIL) >4× the upper limit of normal (ULN) or was deemed unsuitable for trial participation by the investigator; (2) Renal function: serum creatinine >3× upper limit of normal (ULN), urine protein positive and deemed unfit for study; (3) Bone marrow function: absolute value of neutrophil (ANC) <1.0×10^9/L; Platelet (PLT) <20×10^9/L; Hemoglobin (HGB) <70 g/L; (4) Coagulation function: prothrombin time (PT) extended >5s; 7. Persons who have been treated with human plasma preparations (including human blood albumin preparations) within 7 days prior to the initial administration of the experimental drug; People with a history of organ transplantation; Those who need or plan to undergo interventional invasive testing or therapy during the study; 8. Those who have participated in or are participating in clinical trials of other new drugs or medical devices and have used investigational drugs/investigational treatments within 30 days prior to screening; 9. Those who test positive for antibodies to the human immunodeficiency virus (HIV); 10. Pregnant or lactating women; 11. Other reasons why the researcher considered it inappropriate to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Changes in serum albumin concentration | 14 days
  Change in serum albumin concentration from baseline confirmed by albumin examination immediately after completion of last intravenous administration

SECONDARY OUTCOMES:
Ascites depth changes | 57 days
  Change in ascites depth from baseline after administration
Proportion of subjects with serum albumin concentration ≥35 g/L | 14days
  Proportion of subjects with serum albumin concentration ≥35 g/L confirmed by albumin examination at completion of final IV administration
The time when serum albumin concentration reached ≥35 g/L | 57 days
  The time when serum albumin concentration reached ≥35 g/L
Abdominal circumference change | 57 days
  Changes in abdominal circumference from baseline after administration
Weight change | 57 days
  Change in body weight from baseline after administration

CONTACTS AND LOCATIONS:
Overall Officials: dong Ji Jia, Ph.D, Study Director — Beijing Friendship Hospital
Locations (1):
- Shenzhen Protgen Ltd, Guangdong, Shenzhen, China

IPD SHARING:
Plan to Share IPD: No